CLINICAL TRIAL: NCT04685850
Title: Long-term Sequelae of Childhood Meningitis and Meningococcal Purpura Fulminans in Ile de France: a Multidisciplinary Approach
Brief Title: Long-term Sequelae of Childhood Meningitis and Meningococcal Purpura Fulminans
Acronym: SEINE
Status: Terminated | Type: Observational
Why Stopped: lack of inclusion
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Responsible Party: Sponsor
Other Study IDs: SEINE
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Meningitis, Meningococcal; Sequela
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: sequela evaluation — clinical and neurological examination, psychological evaluation (cognitive performance), an auditory, speech and visual assessment and an evaluation of the child's school performance

SUMMARY:
While the initial evolution of meningococcal meningitis (MM) is well described, there are few data on the long-term evolution, beyond 1 year.

The objective of this research is to evaluate the sequelae of MM beyond 1 year in patients with a history of MM followed in Paris area, France. Most children with MM in France have been included in the MM register and are still being followed. Parents will be offered a detailed clinical evaluation of their child including: a clinical and neurological examination, a cognitive performance assessment, an auditory, speech and visual assessment and an evaluation of the child's progress at school.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children from 0 to 17 years old
* Having had meningitis or meningococcal purpura fulminans between 2010 and 2021
* Delay ≥ 1 year between the date of diagnosis of meningitis or purpura meningococcal fulminans and the date of inclusion in the study (signature of the informed consent)
* The holders of parental authority have read and understood the information letter and their express consent has been obtained
* Patient affiliated to a social security system (Social Security or Universal Medical Coverage)

Exclusion Criteria:

* refusal to participate

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from 0 to 17 years old who had meningococcal meningitis between 2010 and 2019
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Number of children with at least one neurological, orthopedic or sensory sequelae | 1 year

SECONDARY OUTCOMES:
Number of children with severe neurological sequelae | 1 year
Number of children with orthopedic complications | 1 year
Number of children with sensory disorders | 1 year
Number of children with skin sequelae | 1 year
Number of children with learning disabilities | 1 year
Number of children with cognitive or psychological difficulties identified on the WPPSI, WISC V or VINELAND depending on their age and capacity | 1 year
  95% of the population has a Total IQ between 70 and 130 (from low intelligence to high intelligence).
Number of consultations during follow-up | 1 year
Post-traumatic stress in parents using the IES-R questionnaire | 1 year
  A score up to 33 is associated with a stress post traumatic

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Bicêtre, Le Kremlin-Bicêtre, Kremlin Bicêtre
  - CHU Annecy, Annecy
  - CHI créteil, Créteil
  - Centre Intercommunal de Villeneuve Saint Georges, Crosne
  - Groupe Hospitalier Nord Essonne, Longjumeau
  - GHEF site de Meaux, Meaux
  - Hôpital Necker Enfants Malades, Paris
  - Robert debré hospital, Paris
  - Ch Pontoise, Pontoise

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baloche A, Jung C, Levy M, Elbez-Rubinstein A, Bechet S, Layouni I, Monguillot G, Taha MK, Cohen R, Levy C. Long-term impact of invasive meningococcal disease in children: SEINE study protocol. PLoS One. 2022 May 26;17(5):e0268536. doi: 10.1371/journal.pone.0268536. eCollection 2022. PMID 35617288
- See also: Long-term impact of invasive meningococcal disease in children: SEINE study protocol — https://pubmed.ncbi.nlm.nih.gov/35617288/